CLINICAL TRIAL: NCT00935207
Title: The Impact of a Pain Diary on the Communication of Pain in Pediatric Patients
Brief Title: Study of the Impact of a Pain Diary in Pediatric Patients
Status: Terminated | Type: Observational
Why Stopped: Poor enrollment and data collection
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Ostrenga, Pharmacist, University of Mississippi Medical Center
Other Study IDs: 2009-0054
Record Dates: First submitted 2009-06-17; First posted 2009-07-08 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Pain
Keywords: Pain; Pediatric Pain; Pain Diary; Pediatric Pain Measurement; Pain Measurement
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Pain Diary: Patients will be give a pain diary to complete.
  Interventions: Other: Pediatric Pain Diary

INTERVENTIONS:
Other: Pediatric Pain Diary — Pain diary designed for pediatric patients

SUMMARY:
The purpose of this study is to show the impact of a pain diary on the communication of pain by pediatric patients. Participants will be given a pain diary after consent and asked to complete the record each time they have pain. A survey about the efficacy of the pain diary will be taken prior to discharge by the nurse, physician, patient and parents. The hypothesis is that the pain diary will improve the communication.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients at the Blair E. Batson Hospital for Children 3-19 years of age, receiving regular controlled substance analgesic defined as: codeine with acetaminophen, fentanyl, hydromorphone, meperidine, morphine, oxycodone with acetaminophen, propoxyphene with acetaminophen, and hydrocodone with acetaminophen.

Exclusion Criteria:

* Admitted to the Pediatric Intensive Care Unit
* Surgical patients, defined as patients having surgery since admission other than minor procedures
* Patients anticipated to receive pain medication for less than 24 hours
* Patients unable to verbally communicate their pain

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Inpatients at the Blair E. Batson Hospital for Children 3-19 years of age, receiving regular controlled substance analgesic defined as: codeine with acetaminophen, fentanyl, hydromorphone, meperidine, morphine, oxycodone with acetaminophen, propoxyphene with acetaminophen, and hydrocodone with acetaminophen.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Child Survey | Hospital discharge
Parent Survey | Hospital Discharge
Nurse Survey | Hospital Discharge
Physician Survey | Hospital Discharge

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ostrenga, Pharm.D., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States